CLINICAL TRIAL: NCT04099628
Title: Diagnostic Tools for Human African Trypanosomiasis Elimination and Clinical Trials: WP3 Post Elimination Monitoring
Acronym: DiTECT-HAT-WP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Ministry of Public Health, Democratic Republic of the Congo (Other Government); Institut National de Sante Publique (Other); CIRDES (Unknown); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Institute of Tropical Medicine, Belgium (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DiTECT-HAT-WP3
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Human African Trypanosomiasis; Sleeping Sickness; Trypanosoma Brucei Gambiense; Infection; West African Sleeping Sickness; African Trypanosomiases; Trypanosomiasis; African, Due to Trypanosoma Brucei Gambiense, Gambiense
Keywords: monitoring; surveillance; re-emergence; rapid diagnostic test; trypanolysis; LAMP; ELISA; molecular biology; RT-PCR; serology; diagnosis; specificity; sensitivity
MeSH Terms: conditions — Trypanosomiasis, African; Infections; Trypanosomiasis; Disease; Hypersensitivity | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Intervention Model Description: Sequential assignement
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic tests (Experimental): Diagnostic tests: Rapid diagnostic test (RDT); Serological and molecular tests on DBS
  Interventions: Diagnostic Test: Rapid diagnostic test (RDT); Serological and molecular tests on DBS

INTERVENTIONS:
Diagnostic Test: Rapid diagnostic test (RDT); Serological and molecular tests on DBS — The population of low to zero prevalence HAT foci will be actively screened for HAT by taking a blood sample for performing 3 rapid diagnostic tests (RDT) and for preparing dried blood spots to perform 4 serological and molecular high throughput reference tests. If at least one of the RDTs, serological or molecular reference tests is positive, parasitological examination is performed twice. The combined results of parasitological examinations serve as reference standard.
  Other Names:
  rHAT Sero-Strip (Coris Bioconcept, Belgium) SD Bioline HAT 1.0 (Standard Diagnostics Korea) HAT Sero-K-Set (Coris Bioconcept, Belgium) Immune trypanolysis: presence of antibodies ELISA: on native LiTat 1.3 + LiTat 1.5 variant surface glycoprotein (VSG) LAMP T. brucei Detection Kit (Eiken) RT-PCR: Trypanozoon 18S, Tbg Trypanosoma gambiense specific glycoprotein (TgsGP)

SUMMARY:
This study determines the feasibility, diagnostic performance and cost for monitoring of eliminated human African trypanosomiasis (HAT) foci using diagnostic algorithms of serological and molecular high throughput tests with and without previous rapid diagnostic test blood screening for early detection of Trypanosoma brucei gambiense HAT re-emergence.

DETAILED DESCRIPTION:
In the last decade, the prevalence of Trypanosoma brucei gambiense (Tbg) human African trypanosomiasis (HAT) has fallen and HAT has been targeted for elimination. At low disease prevalence, HAT control is increasingly integrated into routine activities of peripheral health centres. However, the weak capacity of fixed health structures to implement control activities, lack of coverage, the unspecific clinical picture of HAT, and the existence of asymptomatic cases and animal reservoirs may result in under detection of HAT. To ensure sustainability of zero transmission and to avoid re-emergence caused by remaining Tbg reservoirs, continued post-elimination monitoring is therefore required.

Health workers performing house to house visits in foci with very low HAT prevalence can easily collect blood on filter paper and send it to regional HAT reference centres for analysis. The objective of the DiTECT-HAT-WP3 study is to determine the feasibility and cost of diagnostic algorithms of serological and molecular high-throughput tests on blood on filter paper for post-elimination monitoring, with or without a previous screening with rapid diagnostic tests.

In villages in low to zero prevalence foci in Democratic Republic (DR) Congo, Côte d'Ivoire and Burkina Faso, a health worker will go from house to house to 1) register all consenting inhabitants in a Personal Digital Assistant; 2) take a blood sample on filter paper 3) perform 3 rapid diagnostic tests. All dried blood spots (DBS) are sent to the reference laboratory for high-throughput testing (ELISA, trypanolysis, loop-mediated isothermal amplification method (LAMP) and real time (RT) -PCR). Subjects positive in at least 1 test - the RDTs or high-throughput tests - are revisited twice for parasitological confirmation.

In each country, blood specimens of 6000 persons will be tested. The relative effectiveness and overall cost of the different diagnostic algorithms will be investigated. We will quantify the break-even point for an imperfect test algorithm by formulating a decision criterion to assess how many false negatives, but particularly how many false positives can be tolerated while still achieving an intervention with a reasonable cost burden. The results will enable us to propose a test algorithm and a threshold to send out specialised mobile teams for stopping HAT re-emergence, without unnecessarily raising the alarm.

ELIGIBILITY:
Inclusion Criteria:

* Permanent resident of village (in low to zero prevalence HAT focus) for minimum 1 year

Exclusion Criteria:

* Previously treated for HAT (irrespective of time elapsed since treatment)
* No informed consent
* < 4 years old

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13747 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity for HAT diagnosis of RDT, RDT combinations, algorithms of RDT and serological and/or molecular tests on the population at risk | 6 months
  Index tests: 3 RDTs on fresh blood, immune trypanolysis on DBS, ELISA on DBS, LAMP on DBS, RT-PCR on DBS.
  Reference standard: for index test positives only: combined results of 2 parasitological examinations. Subjects negative in all index tests are considered HAT negative.
Specificity for HAT diagnosis of RDT, RDT combinations, algorithms of RDT and serological and/or molecular tests on the population at risk | 6 months
  Index tests: 3 RDTs on fresh blood, immune trypanolysis on DBS, ELISA on DBS, LAMP on DBS, RT-PCR on DBS.
  Reference standard: for index test positives only: combined results of 2 parasitological examinations. Subjects negative in all index tests are considered HAT negative.

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Lejon, PhD, HDR, Principal Investigator — Institut de Rechercher pour le Développement
Locations (3):
- CIRDES, Bobo-Dioulasso, Burkina Faso
- Institut Pierre Richet, Institut National de Santé Publique, Bouaké, Côte d’Ivoire
- Programme Nationale de Lutte contre la trypanosomiase humaine Africaine, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes